CLINICAL TRIAL: NCT01836900
Title: Endoscopic Treatment of Recurrent Upper GI Bleeding From Gastroduodenal Ulcers: OTSC [Over the Scope Clip] Versus Standard Therapy
Brief Title: Endoscopic Treatment of Recurrent Upper GI Bleeding: OTSC [Over the Scope Clip] Versus Standard Therapy
Acronym: STING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Collaborators: University Hospital Tuebingen (Other); University Hospital Augsburg (Other); Marienkrankenhaus Frankfurt (Other); Klinikum Stadt Hanau (Other); Klinikum Garmisch-Patenkirchen (Other); University of Zurich (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STING
Record Dates: First submitted 2013-04-15; First posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Acute Upper Gastrointestinal Hemorrhage
Keywords: OTSC; Upper gastrointestinal bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Hemostasis, Endoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Therapy (Active Comparator): Endoscopic therapy with Standard Clip + injection of epinephrine solution or thermal therapy + injection of epinephrin-solution
  Interventions: Device: Endoscopic hemostasis
- OTSC (Over The Scope Clip) (Experimental): Endoscopic therapy with Application of OTSC Clip and Injection of epinephrin-solution
  Interventions: Device: Endoscopic hemostasis

INTERVENTIONS:
Device: Endoscopic hemostasis — Hemostasis with Standard Therapy (standard clip or thermal therapy + injection of adrenaline solution) or by application of the Over The Scope Clip and injection of adrenaline solution

SUMMARY:
Prospective-randomized trial. Patients with recurrent bleeding from gastroduodenal ulcers are randomized into either endoscopic treatment with the OTSC [Over The Scope Clip] or endoscopic standard therapy. Hypothesis: Endoscopic therapy with OTSC is superior to standard therapy regarding technical success and rebleeding.

ELIGIBILITY:
Inclusion Criteria:

* Recurrence of bleeding from gastroduodenal ulcers

Exclusion Criteria:

* Malignant ulcers, variceal bleeding, patients younger than 18 years, lesions not suitable for treatment with OTSC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Persistent bleeding or Rebleeding with 7 days | 7 days

SECONDARY OUTCOMES:
blood units transfused | 30 days
duration of hospital stay | 30 days
duration of intensive care unit stay | 30 days
30 d Mortality | 30 days
Amount of endoscopic reinterventions | 7 d
Necessity of surgical or angiographic therapy | 7 d
Complications during or after OTSC (Over The Scope Clip) placement | 7 d

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Germany

REFERENCES:
- [Derived] Schmidt A, Golder S, Goetz M, Meining A, Lau J, von Delius S, Escher M, Hoffmann A, Wiest R, Messmann H, Kratt T, Walter B, Bettinger D, Caca K. Over-the-Scope Clips Are More Effective Than Standard Endoscopic Therapy for Patients With Recurrent Bleeding of Peptic Ulcers. Gastroenterology. 2018 Sep;155(3):674-686.e6. doi: 10.1053/j.gastro.2018.05.037. Epub 2018 May 24. PMID 29803838